CLINICAL TRIAL: NCT00090519
Title: Reduction in the Occurrence of Center-Involved Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8211; B7A-MC-MBDL (Other: Eli Lilly and Company)
Record Dates: First submitted 2004-08-26; First posted 2004-08-31 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — ruboxistaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ruboxistaurin (Experimental): 32 milligrams (mg) once daily (QD) oral for up to 36 months
  Interventions: Drug: ruboxistaurin
- Placebo (Placebo Comparator): QD oral for up to 36 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ruboxistaurin — 32 mg once daily (QD) oral for up to 36 months
  Other Names: LY333531; Arxxant
  Arms: Ruboxistaurin
Drug: placebo — QD oral for up to 36 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if ruboxistaurin can help slow the worsening of an eye disease called macular edema in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes
* 18 years or older
* Non-clinically significant diabetic macular edema
* Mild to moderate diabetic retinopathy in the study eye, vitreous hemorrhage in the study eye
* Relatively good vision (20/30 or better)

Exclusion Criteria:

* Surgery or laser treatment in the study eye
* Glaucoma in the study eye
* Glycosylated hemoglobin (HbA1c) greater than 11%, or systolic blood pressure greater than 170 millimeters of mercury (mmHg)
* Liver disease, dialysis or renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2004-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Beutner, Study Director — Chromaderm, Inc.
Locations (84):
- United States (36):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Artesia, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poway, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Walnut Creek, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New London, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunrise, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wheaton, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peabody, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Independence, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Brunswick, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teaneck, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville Centre, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hershey, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ogden, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parramatta, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sydney, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westmead, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodville, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glostrup Municipality
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sulzbach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- India (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra, Portugal
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valladolid
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District, Taiwan
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool, Merseyside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bristol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Sheetz MJ, Aiello LP, Davis MD, Danis R, Bek T, Cunha-Vaz J, Shahri N, Berg PH; MBDL and MBCU Study Groups. The effect of the oral PKC beta inhibitor ruboxistaurin on vision loss in two phase 3 studies. Invest Ophthalmol Vis Sci. 2013 Mar 11;54(3):1750-7. doi: 10.1167/iovs.12-11055. PMID 23404115
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruboxistaurin | Placebo
Started | 371 | 360
Completed | 298 | 285
Not Completed | 73 | 75
Not completed — Adverse Event | 5 | 4
Not completed — Death | 9 | 9
Not completed — Lost to Follow-up | 26 | 29
Not completed — Withdrawal by Subject | 28 | 29
Not completed — Physician Decision | 2 | 3
Not completed — Sponsor Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruboxistaurin | Placebo | Total
Number analyzed (Participants) | 371 | 360 | 731
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.20 (10.85) | 55.15 (11.18) | 55.17 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 137 | 275
  Male | 233 | 223 | 456
Region of Enrollment [Number; unit: participants]
  United States | 93 | 97 | 190
  Portugal | 15 | 16 | 31
  Taiwan | 3 | 1 | 4
  Spain | 13 | 11 | 24
  Russian Federation | 28 | 24 | 52
  United Kingdom | 21 | 18 | 39
  Italy | 8 | 6 | 14
  India | 25 | 26 | 51
  France | 11 | 10 | 21
  Mexico | 22 | 22 | 44
  Canada | 22 | 25 | 47
  Brazil | 13 | 16 | 29
  Poland | 20 | 16 | 36
  Australia | 20 | 17 | 37
  Denmark | 26 | 28 | 54
  Netherlands | 9 | 8 | 17
  Germany | 22 | 19 | 41
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 29.90 (6.09) | 29.82 (5.89) | 29.86 (5.99)
Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)]
  Systolic Blood Pressure | 132.90 (15.25) | 133.50 (15.58) | 133.20 (5.99)
  Diastolic Blood Pressure | 77.68 (8.68) | 77.77 (9.05) | 77.73 (8.86)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent glycosylated hemoglobin] | 8.14 (1.31) | 8.25 (1.31) | 8.19 (1.31)
Diabetes Type [Number; unit: participants] — Type 1 diabetes results from autoimmune mediated destruction of the beta cells of the pancreas. Participants require insulin treatment to survive. Type 2 diabetes is characterized by resistance to the action of insulin leading to relative insulin deficiency.
  participants
    Type 1 | 85 | 76 | 161
    Type 2 | 286 | 284 | 570
Duration of diabetes [Mean (Standard Deviation); unit: years] | 15.82 (8.00) | 15.57 (7.48) | 15.70 (7.75)
Insulin use [Number; unit: participants]
  Yes | 241 | 228 | 469
  No | 130 | 132 | 262
Number of diabetic retinopathy (DR) study eyes per participant [Number; unit: participants]
  Two | 351 | 336 | 687
  One | 20 | 24 | 44
Visual Acuity Score (Letters Correct) [Mean (Standard Deviation); unit: Letters read correctly] — Visual acuity by the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. Each participant starts at the top of the chart containing 5 letters per row and reads down the chart until reaching a row where a minimum of 3 letters on a line cannot be read. Each participant is scored by how many letters could be correctly identified. A higher number of letters correctly identified represents better visual acuity.
  Letters read correctly | 84.12 (7.93) | 84.27 (7.70) | 84.19 (7.81)
Diabetic Retinopathy (DR) Level [Number; unit: DR study eyes for each level] — DR level is reported by number of DR study eyes for each level (722 DR study eyes in ruboxistaurin group and 696 DR study eyes in placebo group). EDTRS Final Retinopathy Severity Scale ranges from Level 10 (DR absent) to Level 65 (moderate proliferative diabetic retinopathy [PDR]), with a total of 12 levels based on the number of letters read incorrectly. Less than Level 47= mild to moderate nonproliferative diabetic retinopathy (NPDR). Level 47= moderately severe NPDR. Level 53=severe NPDR. Each level represents a change in DR (i.e., a change from Level 47 to >= Level 61 is >=2 steps worse).
  DR study eyes for each level
    <47 | 465 | 421 | 886
    47 | 250 | 272 | 522
    53 | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Duration of Definite Center of Macula-involved Diabetic Macular Edema (DME)
Description: Duration of center of macula involvement when primary study outcome (DME involvement in center of macula determined by central grading of stereoscopic fundus photographs) was identified at a visit, participant was considered to have had definite center involvement for a specified length of time between the adjacent visits. Total duration of center involvement was calculated. Mean duration was total duration of center involvement divided by total number of participants. Participant durations were summarized, total number of months of center involvement in both treatment groups were displayed.
Time Frame: 6 Months through 36 Months
Population: Intent-to-treat (ITT) population including all randomized participants analyzed according to the treatment group to which they were originally assigned by random allocation even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Measure: Mean (Standard Deviation); unit: months per participant
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 349 | 346
months per participant | 1.72 (4.95) | 1.69 (4.41)
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.969, ANOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.714 to 0.686]

2. Secondary Outcome: Change From Baseline in Visual Acuity by Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) Chart at 36 Months
Description: ETDRS VA: participant starts at the top of the chart containing 5 letters per row and reads down the chart until reaching a row where a minimum of 3 letters on a line cannot be read. Participant is scored by how many letters could be correctly identified. A higher number of letters correctly identified represents better visual acuity. Results are reported based on the number of diabetic retinopathy (DR) eyes.
Time Frame: Baseline, 36 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters read correctly
Units Other Than Participants: DR study eyes
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 371 | 360
Number analyzed (DR study eyes) | 722 | 695
Letters read correctly
  Baseline (letters correct) (n=722, 695) | 84.12 (7.93) | 84.27 (7.70)
  Change from baseline (n=687,670) | -1.14 (7.38) | -2.30 (9.21)
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value is for change from baseline; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [0.21 to 1.97]

3. Secondary Outcome: First Occurrence of Focal/Grid Photocoagulation
Description: The first occurrence of focal/grid photocoagulation regardless of diabetic macular edema (DME) distance from the center of the macula.
Time Frame: Baseline through 36 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 371 | 360
participants
  Yes | 32 | 27
  No | 339 | 333
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.577, Chi-squared — P-value is for first occurrence of focal/grid photocoagulation yes versus no

4. Secondary Outcome: Change From Baseline in Contrast Sensitivity by Pelli-Robson
Description: Pelli-Robson chart read from left to right + from top to bottom. Each line has 2 groups, each of 3 letters. Letters in each group have same contrast. Contrast in each successive group is less than the preceding group. Participant reads letters starting with highest contrast, continues until 2 or 3 letters in 1 group are incorrectly named. Scored on key showing all letters at full contrast, gives the log contrast sensitivity corresponding to each group. Score is determined by previous group (last group in which 2 or 3 letters were correctly named). Results reported based on number of DR eyes.
Time Frame: Baseline, 36 Months
Population: Intent-to-treat (ITT) population: all randomized participants analyzed according to treatment group to which they were originally assigned by random allocation even if they did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol.
Measure: Mean (Standard Deviation); unit: Letters read correctly
Units Other Than Participants: DR Study Eyes
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 371 | 360
Number analyzed (DR Study Eyes) | 718 | 689
Letters read correctly
  Baseline (letters correct) (n=718,689) | 33.54 (3.33) | 33.71 (3.54)
  Change from baseline (n=685,664) | -0.54 (3.84) | -1.06 (4.68)
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.041, ANCOVA — P-value is for change from baseline; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.02 to 0.87]

5. Secondary Outcome: Progression of Nonproliferative Diabetic Retinopathy (DR) by Seven-field Stereo Fundus Photography
Description: Participants were classified as having experienced progression or no progression of DR by 36-month visit. Progression of DR=3 steps on ETDRS retinopathy severity person scale for participants with both eyes less than proliferative diabetic retinopathy (PDR) at baseline OR 2 steps on ETDRS retinopathy severity eye scale for participants with 1 eye less than PDR at baseline OR application of panretinal laser therapy. Participants were assigned at baseline to ETDRS retinopathy severity scale for persons or individual eyes; determination of no progression/progression was dependent on the scale.
Time Frame: Baseline through 36 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 371 | 360
participants
  No progression | 328 | 312
  Progression | 43 | 48
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.475, Chi-squared — P-value is for progression of nonproliferative diabetic retinopathy (DR) by seven-field stereo fundus photography progression versus no progression

6. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate
Description: The Modification of Diet in Renal Disease (MDRD) study formula used for the estimated glomerular filtration rate (eGFR) determination is: eGFR = 170 X (Serum creatinine concentration [mg/deciliter (dL)])-0.999 X (Age [years]) -0.176 X (0.762 if participant is female) X (1.180 if participant is black) X (Serum urea nitrogen concentration [mg/dL])-0.170 X (Serum albumin concentration [grams (g)/dL])+0.318.
Time Frame: Baseline, 36 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 square meter
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 368 | 358
milliliter/minute/1.73 square meter
  Baseline (n=368,358) | 85.35 (22.24) | 87.27 (23.44)
  Change from baseline (n=340,328) | -5.55 (15.70) | -7.92 (17.31)
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.211, ANCOVA — P-value is for change from baseline; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [-0.87 to 3.92]

7. Secondary Outcome: Change From Baseline at Endpoint in Albumin/Creatinine Ratio
Time Frame: 36 Months
Population: The completer population includes participants who completed all 36 months of the treatment phase.
Measure: Mean (Standard Deviation); unit: micrograms/millimole (ug/mmol)
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 270 | 261
micrograms/millimole (ug/mmol)
  Baseline (n=270,261) | 123.53 (507.93) | 152.61 (623.98)
  Change from baseline (n=267,253) | 135.90 (865.34) | 72.69 (720.35)
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.365, t-test, 2 sided — P-value is for change from baseline; Mean Difference (Final Values) = 63.22, 95% CI 2-sided [-73.68 to 200.12]

8. Secondary Outcome: Change From Baseline at Endpoint in Visual Function by the National Eye Institute Visual Functioning Questionnaire (NEI VFQ-25) at 36 Months
Description: 25 vision-targeted questions representing 11 vision-related constructs and a 1-item general health rating question. Measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning and task-oriented domains related to daily visual functioning. Each item is converted to a 0 to 100 scale such that a higher score represents better functioning.
Time Frame: 36 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 351 | 342
units on a scale
  Baseline (n=351,342) | 67.86 (8.25) | 67.56 (7.85)
  Change from baseline (n=314,309) | 0.17 (6.21) | -1.36 (8.56)
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value is for change from baseline; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [0.38 to 2.66]

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Summaries of serious adverse events (SAEs) and all other non-serious adverse events (AEs) are located in the Reported Adverse Event Module.
Time Frame: Baseline through 36 Months
Population: Safety population: all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 371 | 360
participants
  Serious adverse events | 93 | 82
  Adverse events | 298 | 299

10. Primary Outcome: Occurrence of Sustained Moderate Visual Loss (SMVL) in a Diabetic Retinopathy (DR) Study Eye
Description: The occurrence of SMVL was defined as ≥15 letter decrease from baseline in best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) in any DR study eye relative to baseline that is sustained for the last 6 months of participation. ETDRS VA: participant starts at the top of the chart containing 5 letters per row and reads down the chart until reaching a row where a minimum of 3 letters on a line cannot be read. Participant is scored by how many letters could be correctly identified. A higher number of letters correctly identified represents better visual acuity.
Time Frame: Baseline, 36 Months
Population: Intent-to-treat (ITT) population: all randomized participants with at least 1 eligible study eye analyzed according to the treatment group to which they were originally assigned by random allocation even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 342 | 331
participants
  Yes | 8 | 16
  No | 334 | 315
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.081, Chi-squared — P-value is for occurrence of sustained moderate visual loss (SMVL) in a diabetic retinopathy (DR) study eye yes versus no; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.20 to 1.12]

ADVERSE EVENTS:
Arm/Group | Ruboxistaurin | Placebo
Serious Adverse Events (participants affected / at risk) | 93/371 | 82/360
Other Adverse Events (participants affected / at risk) | 298/371 | 299/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruboxistaurin (N=371) | Placebo (N=360)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (3) | 5 (5)
Angina pectoris (Cardiac disorders) | 4 (14) | 1 (1)
Angina unstable (Cardiac disorders) | 3 (4) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (10) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (5) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (4) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (8)
Cardiac failure congestive (Cardiac disorders) | 1 (4) | 2 (9)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (4) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (9) | 5 (16)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 6 (6) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (11)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 1 (8) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (7)
Ocular myasthenia (Eye disorders) | 1 (4) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Calcinosis (General disorders) | 1 (3) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (2)
Chest pain (General disorders) | 3 (3) | 1 (1)
Death (General disorders) | 0 (0) | 3 (3)
Impaired healing (General disorders) | 0 (0) | 1 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (2) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (6) | 0 (0)
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 (9) | 6 (6)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 2 (7)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (10) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (10) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (11)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (14) | 0 (0)
Angioimmunoblastic t-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (4)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (5)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (4) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (4) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (7) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (5) | 2 (3)
Coma hepatic (Nervous system disorders) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (9) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (7) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (5)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (12) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (4) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 2 (7) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (9)
Renal artery arteriosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (11) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (4) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (4) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (4) | 2 (15)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (4)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Splenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (13) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (4) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 2 (11) | 2 (5)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruboxistaurin (N=371) | Placebo (N=360)
Diarrhoea (Gastrointestinal disorders) | 38 (90) | 32 (108)
Nausea (Gastrointestinal disorders) | 17 (23) | 21 (60)
Vomiting (Gastrointestinal disorders) | 19 (22) | 17 (25)
Oedema peripheral (General disorders) | 16 (60) | 24 (86)
Pyrexia (General disorders) | 15 (18) | 19 (19)
Bronchitis (Infections and infestations) | 19 (28) | 16 (23)
Influenza (Infections and infestations) | 47 (67) | 36 (58)
Nasopharyngitis (Infections and infestations) | 65 (135) | 59 (121)
Sinusitis (Infections and infestations) | 24 (54) | 13 (20)
Upper respiratory tract infection (Infections and infestations) | 17 (25) | 20 (34)
Urinary tract infection (Infections and infestations) | 20 (42) | 18 (40)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 28 (129) | 29 (131)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (89) | 35 (144)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (93) | 36 (105)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (56) | 24 (83)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 (82) | 22 (99)
Headache (Nervous system disorders) | 37 (102) | 44 (129)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (73) | 46 (85)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 (36) | 24 (36)
Hypertension (Vascular disorders) | 43 (229) | 49 (282)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days